CLINICAL TRIAL: NCT04372238
Title: The Rhode Island Prescription and Illicit Drug Study Responding to Fentanyl and Associated Harms
Brief Title: The Rhode Island Prescription and Illicit Drug Study
Acronym: RAPIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1904002388; R01DA047975 (NIH)
Record Dates: First submitted 2020-03-02; First posted 2020-05-01 (Actual); Results first posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-07

CONDITIONS: Opioid Overdose; Drug Overdose
Keywords: Drug overdose; Substance-Related Disorders; Chemically-induced disorders; Fentanyl; analgesics, Opioids; Narcotics; Naloxone; Central Nervous System Depressants; Physiological Effects of Drugs
MeSH Terms: conditions — Opiate Overdose; Drug Overdose; Substance-Related Disorders; Chemically-Induced Disorders

STUDY DESIGN:
Intervention Model Description: Participants randomized to receive the RAPIDS intervention will receive fentanyl test strips and additional fentanyl-specific education. Both arms will receive standardized overdose prevention education and naloxone.
Who Masked: Outcomes Assessor
Masking Description: The biostatistician will be blinded to the intervention/control group assignment throughout the course of the study and the assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RAPIDS intervention (Experimental): Participants randomized to receive the RAPIDS intervention will receive a fentanyl specific behavioral intervention and a brief behavioral intervention to increase willingness to use fentanyl test strips and engage in overdose risk reduction behaviors, in addition to standard OEND.
  Interventions: Behavioral: RAPIDS Intervention; Behavioral: Standard OEND
- Standard OEND (Active Comparator): In the control arm participants will receive standard overdose education and naloxone distribution (OEND).
  Interventions: Behavioral: Standard OEND

INTERVENTIONS:
Behavioral: RAPIDS Intervention — RAPIDS intervention combines a behavioral intervention along with hands-on training to use fentanyl test strips.
  Arms: RAPIDS intervention
Behavioral: Standard OEND — In the attention-matched control arm, participants will receive standardized overdose education and naloxone distribution (OEND) training, with attention-control visits at 1, 2, and 3 months. Participants will receive a naloxone kit after completion of the first session, and information regarding where to obtain additional naloxone at subsequent visits. They will have contact with study staff at month 6 and 12 follow-up visits to capture outcome and covariate data.

SUMMARY:
This study will test the efficacy of a novel drug-checking intervention to prevent fatal and non-fatal overdose among people who use drugs (PWUD), who are 18-65 years old at the time of enrollment. The investigators will evaluate whether the incorporation of rapid fentanyl testing into a theory-driven overdose education and prevention intervention reduces rates of overdose compared to standard overdose education and naloxone distribution. Results from this study will significantly improve public health efforts to address the fentanyl overdose epidemic and reduce harms associated with exposure to drugs contaminated with fentanyl. This is a full clinical trial, building on the previously approved fentanyl-test-strip pilot study (2016-2017), the results of which have recently been published.(Krieger et al., 2018)

DETAILED DESCRIPTION:
The investigators will assess the efficacy of the RAPIDS intervention on preventing overdose among PWUD. Participants will be randomized 1:1 to receive the RAPIDS intervention or the attention-matched control condition. Experimental arm participants will receive the RAPIDS intervention, which includes education about the dangers of illicitly manufactured fentanyl (IMF), motivational interviewing to increase willingness to use fentanyl test strips and engage in overdose risk reduction behaviors, hands-on training to use the test strips, and opportunities to plan and role- play how to implement overdose risk reduction behaviors upon receipt of a positive or negative test result. In the attention-matched control arm, participants will receive standardized overdose education and naloxone distribution (OEND) training. All participants will attend additional study visits at months 1,2,3,6, and 12. The primary endpoint will be the rate of self-reported overdose over the follow-up period. Secondary endpoints (e.g., overdose death) will be ascertained by data linkage to statewide overdose surveillance databases.

The primary aims of this study are to: 1) Assess the efficacy of the RAPIDS intervention in reducing rates of overdose among people who use drugs; 2) Examine the degree to which reductions in rates of overdose are mediated by increases in information, motivation, behavioral skills, and self-efficacy regarding fentanyl, rapid fentanyl testing, and harm reduction practices; and 3) Explore whether there is heterogeneity of treatment effect related to key participant characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Reside in Rhode Island
* Are able to complete interviews in English
* Are able to provide informed consent
* Self-report past 30 day heroin, illicit stimulants, counterfeit prescription pills, or injection drugs

Exclusion Criteria:

* Participants who exclusively misuse medications obtained from a physician or diversion from someone else's prescription

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 509 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brandon DL Marshall, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University School of Public Health, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krieger MS, Goedel WC, Buxton JA, Lysyshyn M, Bernstein E, Sherman SG, Rich JD, Hadland SE, Green TC, Marshall BDL. Use of rapid fentanyl test strips among young adults who use drugs. Int J Drug Policy. 2018 Nov;61:52-58. doi: 10.1016/j.drugpo.2018.09.009. Epub 2018 Oct 18. PMID 30344005
- [Derived] Jacka BP, Goldman JE, Yedinak JL, Bernstein E, Hadland SE, Buxton JA, Sherman SG, Biello KB, Marshall BDL. A randomized clinical trial of a theory-based fentanyl overdose education and fentanyl test strip distribution intervention to reduce rates of opioid overdose: study protocol for a randomized controlled trial. Trials. 2020 Nov 26;21(1):976. doi: 10.1186/s13063-020-04898-8. PMID 33243291

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through flyers, bus advertisements, through word of mouth or directly from syringe services providers. Study visits happened at three locations, two of which were drop in sites within syringe services programs and the other was our study office.
Pre-assignment Details: There were a number of participants who left during the baseline visits, largely due to needing to get to another appointment, and therefore did not receive allocation.
Period: Overall Study
Arm/Group | RAPIDS Intervention | Standard OEND
Started | 254 | 255
Completed | 245 | 242
Not Completed | 9 | 13
Not completed — Duplicate | 3 | 3
Not completed — Did not consent for data linkage | 6 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RAPIDS Intervention | Standard OEND | Total
Number analyzed (Participants) | 245 | 242 | 487
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 41 [35 to 52] | 44 [34 to 54] | 43 [35 to 53]
Sex: Female, Male [Count of Participants; unit: Participants] — Not all of our participants reported sex. Some preferred to not answer the question. Population: A number of our participants refused to answer this question in a way presented in the table below
  Participants
    number analyzed (Participants) | 243 | 233 | 476
    Female | 81 | 85 | 166
    Male | 162 | 148 | 310
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 135 | 116 | 251
  Non-Hispanic Black | 33 | 44 | 77
  Non-Hispanic Multiracial | 29 | 26 | 55
  Hispanic/Latine | 47 | 55 | 102
  Unknown | 1 | 1 | 2
Self-reported non fatal overdose [Count of Participants; unit: Participants] | 15 | 12 | 27
One or more EMS runs for suspected opioid overdose [Count of Participants; unit: Participants] | 22 | 27 | 49
One or more emergency department encounters for non-fatal overdose [Count of Participants; unit: Participants] | 18 | 28 | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of People Identified Has Having One or More Overdose Among RAPIDS Trial Participants
Description: A composite measure was created in order to be able to create a count of overdoses experienced at 6 or 12 months post baseline. This was from a combination of sefl-reported data, and administrative data.
Time Frame: 12 months post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | RAPIDS Intervention | Standard OEND
Number analyzed (Participants) | 245 | 242
Participants | 48 | 36

2. Primary Outcome: Accidental Non-fatal Overdose in the Past Month
Description: At each visit, we asked participants a yes or no question as to whether they experienced an overdose in the last month. This self-reported outcome was creating by taking the number of people who reported an overdose at a given time increment and dividing it by the total number of visits completed at that time increment. We did this for each arm. So for example, at month 1, the calculation would have been
  [number of intervention participants reporting an overdose at baseline]/[total visits completed by intervention participants at month 1]
Time Frame: 12 months post-randomization
Measure: Number; unit: Overdoses per 100 study visits
Arm/Group | RAPIDS Intervention | Standard OEND
Number analyzed (Participants) | 245 | 242
Overdoses per 100 study visits
  Month 1 | 5.4 | 2.7
  Month 2 | 5.6 | 4.6
  Month 3 | 3.4 | 4.0
  Month 6 | 10.6 | 4.3
  Month 12 | 5.3 | 11.7

3. Secondary Outcome: The Number of Fatal Overdose Events
Description: The number of fatal overdoses experienced throughout 12 month enrollment in the study, measured using Rhode Island Department of Health data
Time Frame: 12 months post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | RAPIDS Intervention | Standard OEND
Number analyzed (Participants) | 245 | 242
Participants | 9 | 7

4. Secondary Outcome: Number of Participants With Positive Dry Blood Spot Samples
Description: As part of the dry blood spot supplement, we gathered dry blood spots from participants at baseline and 6 and 12 months post randomization. This outcome assess how many participants in each arm had a positive fentanyl sample.
  Because of protocols at Brown University related to biosafety, we were only able to collect dry blood spots from participants who we met with at our study offices. We could not get samples from those who we recruited from SSPs
Time Frame: 12 months post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | RAPIDS Intervention | Standard OEND
Number analyzed (Participants) | 245 | 242
Participants
  Positive | 34 | 35
  Negative | 86 | 79
  Not assessed | 125 | 128

ADVERSE EVENTS:
Time Frame: Each participant was assessed for all adverse events at an on-going basis for up to 15 months following enrollment.
Description: Severe adverse event data were reported to the IRB and DSMB within 48 hours of occurring, and non-severe adverse events were reported annually.
Arm/Group | RAPIDS Intervention | Standard OEND
All-Cause Mortality (participants affected / at risk) | 9/245 | 7/242
Serious Adverse Events (participants affected / at risk) | 15/245 | 12/242
Other Adverse Events (participants affected / at risk) | 0/245 | 0/242
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAPIDS Intervention (N=245) | Standard OEND (N=242)
Non-fatal overdose (Injury, poisoning and procedural complications) | 15 (15) | 12 (245) — All self-reported non-fatal overdoses were considered to be sever adverse events for this trial

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/38/NCT04372238/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-24): https://cdn.clinicaltrials.gov/large-docs/38/NCT04372238/SAP_001.pdf
  • Informed Consent Form (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/38/NCT04372238/ICF_002.pdf